CLINICAL TRIAL: NCT04394338
Title: The Plastic Covering Method for Self-gripping Mesh Placement in Laparoscopic Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MURA2020/184
Record Dates: First submitted 2020-05-07; First posted 2020-05-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Laparoscopic Inguinal Hernia Repair
Keywords: inguinal hernia repair; laparoscopic inguinal hernia repair; self-gripping mesh placement

STUDY DESIGN:
Intervention Model Description: A randomized control trail comparing the duration of mesh placement and surgeon satisfaction of self-gripping mesh with plastic sheath and with non-plastic sheath covering mesh. Patients with groin hernia who planned for elective laparoscopically repair hernia with self-gripping mesh at Ramathibodi Hospital, Faculty of Medicine, Mahidol University will are informed of the details of research at the outpatient department before admission. 1:1 open label randomization trail was designed dividing the patients into two groups by the study number. The operation will be done with the standard laparoscopic hernia repair technique by experienced surgeons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plastic sheath covering (Active Comparator): plastic sheath was prepared with the standard 9 cmx15cm self-gripping mesh. Then the meshe were folded and unfolded over or under the plastic sheaths in different directions.
  Interventions: Other: self-gripping mesh placement with plastic sheath in laparoscopic inguinal hernia
- mesh placement without plastic sheath (No Intervention): self-gripping mesh were placed without plastic sheath.

INTERVENTIONS:
Other: self-gripping mesh placement with plastic sheath in laparoscopic inguinal hernia — to apply these to the mesh graft placement process. In the first step, plastic sheaths self-gripping mesh placement with plastic sheathwere prepared configuration with the standard 9cmx15cm self-gripping mesh. Then the meshes were folded and unfolded over or under the plastic sheaths.
  Arms: plastic sheath covering

SUMMARY:
Inguinal hernia is one of the most-common surgical conditions. Incidence is about 27% in males and 3% in females.The treatment of this condition is inguinal hernia repair operation which can be approached with several techniques; open hernia repair, laparoscopic hernia repair and robotic hernia repair. The current guidelines recommend the hernia repair operation with mesh placement either Lichtenstenstein operation or laparoscopic technique; transabdominal preperitoneal technique (TAPP) and totally extraperitoneal technique (TEP). In the laparoscopic approach, one of the complications that can occur is post-operative pain from the mesh fixator. So the self-gripping mesh becomes another option to decrease this incidence.However the adhesive property of the mesh is still challenging for many surgeons. Several techniques of self-gripping mesh placement were introduced. One of the popular techniques is bilateral vertical folding of self-gripping mesh which still causes some adhesive problems when introduced to the target area. This research's aim is to present a new technique of the self-gripping mesh placement which is more effective, more convenient, and decreases the time taken to place the mesh at the surgery site.

DETAILED DESCRIPTION:
A randomized control trail comparing the duration of mesh placement and surgeon satisfaction of self-gripping mesh with plastic sheath and with non-plastic sheath covering mesh. Patients with groin hernia who planned for elective laparoscopically repair hernia with self-gripping mesh at Ramathibodi Hospital, Faculty of Medicine, Mahidol University will are informed of the details of research at the outpatient department before admission. 1:1 open label randomization trail was designed dividing the patients into two groups by the study number. The operation will be done with the standard laparoscopic hernia repair technique by experienced surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic inguinal hernia repair

Exclusion Criteria:

* Rejected or withdrawn consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Duration | 5 min
  the duration of self-gripping mesh placement with plastic sheath

SECONDARY OUTCOMES:
post operative pain: pain scores | 24 hours after surgery
  During a preoperative visit, the patients are introduced to the concept of the visual analogue scale (VAS), which ranges from 0 = no pain to 10 = worst pain. The measure pain scores (Visual Analog Scale) in the postoperative period.
wound infection | 30 days
  wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital, Mahidol University
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No